CLINICAL TRIAL: NCT00541502
Title: A Obervational, Prospective Study to Evaluate the Effectiveness of Improving Cognitive Function of Aripiprazole in Treating Adolescents and Young Adults With Psychotic Disorder in Taiwan
Brief Title: Improving Cognitive Function of Aripiprazole in Treating Adolescents and Young Adults With Psychotic Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 31-06-P04
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Psychotic Disorders
Keywords: evaluate the effectiveness of improving cognitive function of aripiprazole in treating adolescents and young adults with psychotic disorder in Taiwan
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a 24-week, observational, prospective study to evaluate the effectiveness of improving cognitive function of aripiprazole in treating adolescents and young adults with psychotic disorder in Taiwan. Approximately 120 qualified patients who have clinical diagnosis of DSM-IV of psychotic symptom (e.g. schizophrenia or other psychotic disorders such as schizophreniform disorder, schizoaffective disorder, delusional disorder, shared psychotic disorder, bipolar disorder with psychotic feature or psychotic disorder not otherwise specified.) will be recruited to achieve at least 100 evaluable subjects. After signing the informed consent form, the demographics, medical history and concomitant medication will be recorded. Besides, physical examination, vital sign, BMI, DSM-IV multiaxial examination, CGI-S and menstrual history will be conducted. Laboratory tests and pregnancy test will be optionally conducted. After evaluating all variables obtained, the eligible patients will be enrolled into study. Patients who fulfill the inclusion / exclusion criteria will be performed the CPT, WCST, BPRS and WHOQOL. Afterwards, patients will be given their first medication at this visit (5 mg ~ 30 mg daily by subject). Besides, the switching period is maximum 8 weeks and is depended upon the clinical judgment of investigator. Efficacy will be evaluated by the change from baseline in Continuous Performance Test (CPT), Wisconsin Card Sorting Test (WCST), Clinical Global Impression Scale (CGI), Brief Psychiatric Rating Scale (BPRS) and The World Health Organization Quality of Life questionnaire (WHOQOL). Safety will be evaluated by the frequency of adverse events, abnormal laboratory results, physical examination, vital sign, BMI and menstrual history for female subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in age between 12 and 25 years old.
2. Clinical diagnosis of DSM-IV of psychotic symptom (e.g. schizophrenia or other psychotic disorders such as schizophreniform disorder, schizoaffective disorder, delusional disorder, shared psychotic disorder, bipolar disorder with psychotic feature or psychotic disorder not otherwise specified.).
3. CGI-S ≧ 3 at screening visit.
4. Informed Consent was obtained from the subject (and legal guardian as if necessary).

Exclusion Criteria:

1. Pregnant or breast feeding women or planning a pregnancy.
2. Patient received electroconvulsive therapy within 4 weeks before the screening visit.
3. Patient has a history of hypersensitivity or allergy to investigated drug.
4. A known severe adverse event related to any antipsychotic medication (including but not limited to haloperidol, chlorpromazine, thioridazine, pimozide, risperidone, quetiapine, ziprasidone).
5. Any clinical condition or significant concurrent disease judged by the investigator to complicate the evaluation of the study treatment.

Ages: 12 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Dates: Start 2007-11; Study Completion 2008-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chih-Ken, PhD, Principal Investigator — Chang Gung Memorial Hospital, Keelung, Taiwan